CLINICAL TRIAL: NCT01792310
Title: A Phase 1/2A Dose Escalation Study of LAM561 in Adult Patients With Advanced Solid Tumours Including Malignant Glioma
Brief Title: A Phase 1/2A Study of LAM561 in Adult Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Laminar Pharmaceuticals (Industry)
Collaborators: Specialized Medical Services (SMS)-Oncology BV (Unknown); Royal Marsden NHS Foundation Trust (Other); Northern Institute for Cancer Research, Newcastle (Unknown); Vall d'Hebron Institute of Oncology (Other); Instituto Oncológico IMQ, Clínica IMQ Zorrotzaurre. Bilbao (Unknown); Onkologikoa, San Sebastián. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIN-001-1203; EudraCT 2012-001527-13 (Registry Identifier: EudraCT NUMBER: 2012-001527-13)
Record Dates: First submitted 2012-12-24; First posted 2013-02-15 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Glioma; Other Solid Tumours
Keywords: Glioma; Solid Tumours; LAM561
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Dose Cohort 1 (Experimental): Intervention: LAM561. 7 dose cohorts of up to 6 patients have been performed in the dose escalation phase. The starting dose cohort received 250 mg twice daily.
  Interventions: Drug: LAM561
- Dose Cohort 2 (Experimental): Intervention: LAM561. 500 mg twice daily
  Interventions: Drug: LAM561
- Dose Cohort 3 (Experimental): Intervention: LAM561.
  1g twice daily
  Interventions: Drug: LAM561
- LAM561 Dose Cohort 4 (Experimental): Intervention: LAM561. 2g twice daily
  Interventions: Drug: LAM561
- LAM561 Dose Cohort 5 (Experimental): Intervention: LAM561. 4g twice daily
  Interventions: Drug: LAM561
- LAM561Dose Cohort 6 (Experimental): Intervention: LAM561. 4g three times daily
  Interventions: Drug: LAM561
- LAM561 Dose Cohort 7 (Experimental): Intervention: LAM561. 8g twice daily
  Interventions: Drug: LAM561
- LAM561 Dose Expansion cohort. Glioma (Experimental): Intervention: LAM561 at the MTD: 4g three times daily. Up to 10 patients with malignant glioma.
  Interventions: Drug: LAM561
- LAM561 Dose Expansion cohort. Non-glioma (Experimental): Intervention: LAM561 at the MTD: 4g three times daily. Up to 10 patients with other advanced solid tumours that are suitable for biopsy.
  Interventions: Drug: LAM561

INTERVENTIONS:
Drug: LAM561 — Patients will receive treatment cycles of 21 days, until any criterion for discontinuation (clinical or radiological progression of disease, clinically unacceptable toxicity, or another "general" discontinuation criterion) is met.
  Patients are expected to receive between one and 6 cycles of treatment. The treatment period may be extended if clinical benefit is shown.
  In the event of significant GI toxicity, the treatment schedule may be modified from continuous dosing to an intermittent regime In the case of toxicity, the dose of LAM561 may be reduced or delayed by up to 14 days at the discretion of the Investigator. A maximum of two dose reductions will be permitted per patient. Treatment "holidays" of no more than 14 days are also permitted for reasons other than toxicity. Intra-patient dose escalation may be permitted in certain specific circumstances.

SUMMARY:
This is a phase 1/2A, open label, non-randomized study in patients with advanced solid tumours including malignant glioma

DETAILED DESCRIPTION:
This is an open label, non-randomized study in patients with advanced solid tumours including malignant glioma. The study will be performed in two phases - a dose escalation phase following a standard "3+3" design to establish dose-limiting toxicity (DLT) and a safe dose of LAM561 followed by two expanded safety cohorts (approximately 10 of whom have malignant glioma and approximately 10 of whom have other advanced solid tumours that are suitable for biopsy) treated at the maximum tolerated dose (MTD). If the MTD is well tolerated in the expanded safety cohorts, that dose becomes the recommended phase 2 dose (RP2D). During each dose cohort, at least one week must elapse between the first and subsequent patients receiving treatment with LAM561. Patients may receive palliative localized radiotherapy, if needed (however, this lesion cannot be a target lesion for evaluation of the treatment response).

Safety, pharmacokinetics (PK), pharmacodynamics and efficacy will be evaluated during the study at pre-defined timepoints

ELIGIBILITY:
Inclusion Criteria

* Males or females providing written, informed consent
* Histologically- or cytologically-confirmed advanced solid malignancy that is refractory to standard-of-care treatment, or for which there is no standard therapy. If this is glioma:Grade III / Grade IV malignant glioma recurring or progressing after first or second line standard-of-care treatment and true progressive disease, confirmed according to the RANO criteria 4.
* Life-expectancy of at least 12 weeks
* Eastern cooperative oncology group (ECOG) performance status of 0-2
* Safety laboratory tests and ECGs within specified limits.
* Using adequate contraception, where applicable
* Presence of lesions suitable for biopsy (mandatory for non-glioma patients enrolled in the expanded safety cohort and highly desirable for non-glioma patients enrolled in the dose escalation phase)

Exclusion Criteria

* Anti cancer therapy within 4 weeks (6 weeks for mitomycin and nitrosureas and 2 weeks for palliative radiotherapy)
* NCI Common terminology criteria for adverse events (CTCAE) >Grade 1 toxicities from prior chemotherapy or radiotherapy that could impact on safety outcome assessment
* Recent >Grade 1 intracranial or intratumoural haemorrhage either by CT or MRI scan. Patients with resolving haemorrhage changes, punctuate haemorrhage or haemosiderin may enter the study
* Significant or uncontrolled cardiovascular disease, unstable angina or myocardial infarction within the preceding 6 months
* Known impairment of GI function that could alter the absorption of study drug
* History of uncontrolled hyperlipidemia and/or the need for concurrent lipid lowering therapy
* Concurrent severe and/or uncontrolled other medical disease that could compromise participation in the study
* Taking warfarin, phenytoin or sulphonylureas (glibenclamide, glimepiride, glipizide, glyburide or nateglanide)
* Pregnant or breast feeding Other protocol specific criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | From the first dose of study drug until 30 days after the last dose of study drug
  All adverse events will be recorded including clinically significant physical examinations and vital signs, laboratory safety tests and 12-lead electrocardiograms

SECONDARY OUTCOMES:
Concentration of LAM561 in blood measured by LC-MS/MS | 21 days
  Full profiles on Day 1 and Day 21 (dose escalation phase only), trough measurements on Day 8, 15 and 21
Concentration of biomarkers in blood or tumour tissue | First 22 days then every 9 cycles until any criterion for discontinuation is met (clinical or radiological progression of disease, clinically unacceptable toxicity, or another "general" discontinuation criterion)
  Effect on glial fibrillary acidic protein in glioma patients and effect on sphingomyelin and dihydrofolate reductase in patients with other solid tumours
Concentration of micro RNA in blood | First 22 days then every 9 cycles until any criterion for discontinuation is met (clinical or radiological progression of disease, clinically unacceptable toxicity, or another "general" discontinuation criterion)
  Blood samples for future analysis of micro RNA
Radiological disease progression | Every 6 weeks until any criterion for discontinuation is met (clinical or radiological progression of disease, clinically unacceptable toxicity, or another "general" discontinuation criterion)
  Measurement by CT or MRI scan. Changes scored according to Response Assessment in Neuro-oncology (RANO) criteria (for glioma patients) or Response evaluation criteria in solid tumours (RECIST v1.1) (for other solid tumour patients).
Clinical disease progression | until any criterion for discontinuation is met (clinical or radiological progression of disease, clinically unacceptable toxicity, or another "general" discontinuation criterion

CONTACTS AND LOCATIONS:
Overall Officials: Professor Johann de Bono, MB ChB FRCP MSc PhD, Study Chair — The Institute of Cancer Research, 15 Cotswold Road, Belmont, Sutton, Surrey, United Kingdom SM2 5NG; Prof. Ruth Plummer, BMBCh, MRCP, Cert Me, Principal Investigator — Northern Institute for Cancer Research, Newcastle; Dr Jordi Rodon, Principal Investigator — Vall d'Hebron Institute of Oncology; Dr Juanita Lopez, Principal Investigator — The Institute of Cancer Research, 15 Cotswold Road, Belmont, Sutton, Surrey, United Kingdom SM2 5NG; Dr Ricardo Fernandez Rodriguez, Principal Investigator — Instituto Oncológico IMQ, Clínica IMQ Zorrotzaurre. Bilbao; Dr Ander Urruticoechea Ribate, Principal Investigator — Onkologikoa, San Sebastián.
Locations (5):
- Spain (3):
  - Vall D'Hebron Institute of Oncology, Barcelona
  - Instituto Oncológico IMQ, Clínica IMQ Zorrotzaurre, Bilbao
  - Onkologikoa, San Sebastián
- United Kingdom (2):
  - Sir Bobby Robson Cancer Trials Research Centre, The Northern Centre for Cancer Care, Freeman Hospital, Newcastle, Newcastle Upon Tyne
  - The Royal Marsden Hospital Drug Development Unit, Sutton, Surrey

REFERENCES:
- [Derived] Lopez J, Lai-Kwon J, Molife R, Welsh L, Tunariu N, Roda D, Fernandez-Garcia P, Llado V, McNicholl AG, Rossello CA, Taylor RJ, Azaro A, Rodon J, Sludden J, Veal GJ, Plummer R, Urruticoechea A, Lahuerta A, Mujika K, Escriba PV. A Phase 1/2A trial of idroxioleic acid: first-in-class sphingolipid regulator and glioma cell autophagy inducer with antitumor activity in refractory glioma. Br J Cancer. 2023 Sep;129(5):811-818. doi: 10.1038/s41416-023-02356-1. Epub 2023 Jul 24. PMID 37488446